CLINICAL TRIAL: NCT03985566
Title: Effects of Fixed Meals With Special Formulated Rice on Blood Glucose Levels of Healthy Volunteers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Alchemy Foodtech Pte Ltd (Unknown)
Responsible Party: Principal Investigator, Mei Hui Liu, Principal Investigator, National University of Singapore
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2017/01126
Record Dates: First submitted 2019-06-10; First posted 2019-06-13 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This study is a within-subject cross-over trial design to assess the glycemic response of fibre enriched rice consumer by human subjects as compared to normal non-enriched rice in a mixed meal setting.
Who Masked: Participant
Masking Description: Fibre Grains have similar appearance to normal Jasmine white rice. It is made up of functional fibre extruded into grain-shaped food particles .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibre Grains (Experimental): Fibre grains were used to partially replaced Jasmine white rice in this arm.
  Interventions: Dietary Supplement: Fibre Grain
- Jasmine white rice (Placebo Comparator): Jasmine white rice is used as a control to compare the outcome.
  Interventions: Dietary Supplement: Jasmine white rice

INTERVENTIONS:
Dietary Supplement: Fibre Grain — Healthy subjects will be provided with 30% Fibre Grain in a mixed meal. After consumption of the meal, the glucose and insulin response will be compared.
  Arms: Fibre Grains
Dietary Supplement: Jasmine white rice — Healthy subjects will be provided with Jasmine white rice in a mixed meal. After consumption of the meal, the glucose and insulin response will be compared.
  Arms: Jasmine white rice

SUMMARY:
The aim of the study is to compare Diabetec® Fibre Grains (FIbre Grains) in a mixed meal setting with Jasmine rice. This is to see whether partial replacement of white rice with Fibre Grains can reduce postprandial blood glucose control.

DETAILED DESCRIPTION:
Lifestyle modification, in particular adopting an appropriate dietary pattern, is generally accepted as the cornerstone for the treatment of people with type 2 diabetes. Consumption of low GI food has shown to improve glycemic control, lipid profile and reduce systemic inflammation. However, there are few dietary intervention studies attempting to change the GI of food by changing the staple carbohydrates. In this study, formulated rice with special fibre enrichment, Fibre Grains, was used to replace rice as the staple carbohydrates in one's diet. This fibre enriched rice has been previously tested to have a lower GI than normal rice while still able to preserve all the sensory characteristics of normal rice. With rice being a staple to Asians, this specially formulated fibre enriched rice offers a lower GI alternative to the conventional rice without affecting the people dietary preference.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Age between 21-65 years old
* Overtly healthy males or females, as determined by medical history, physical examination and laboratory results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator.
* Males and females with stable medical problems that, in the investigator's opinion, will not significantly alter the performance of the biomarker panel, will not place the subject at increased risk by participating in the study, and will not interfere with interpretation of the data.
* Not on any regular medications (western / traditional medicine). Nutritional supplements with established chemical composition that can be ascertained and clearly recorded is acceptable. However, subjects using traditional medicine (with compositions that cannot be ascertained) will be excluded in this study
* Have venous access sufficient to allow for blood sampling as per the protocol
* Reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Family history of diabetes (Parents and/or grandparents with history of diabetes).

Exclusion Criteria:

* History or presence of current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, malignancy or neurological disorders capable of significantly altering the performance of the biomarker panel; or of interfering with the interpretation of data
* Known or ongoing psychiatric disorders within 3 years
* Regularly use known drugs of abuse within 3 years
* Women who are pregnant or lactating
* Have donated blood of more than 500 mL within 4 weeks of study enrolment
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females):• 1 unit = 12 oz or 360 mL of beer; • 5 oz or 150 mL of wine; • 1.5 oz or 45 mL of distilled spirits
* Uncontrolled hypertension (blood pressure [BP] >160/100mmHg
* Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 19 Treatment with any investigational drug, or biological agent within one (1) month of screening or plans to enter into an investigational drug/ biological agent study during the duration of this study
* Known allergy to insulin
* History of bleeding diathesis or coagulopathy
* Any of the following laboratory values at screening:Fasting glucose >=126mg/dL(>=7mmol/L) or 2 hour post-prandial glucose >=200mg/dL (>=11.1mmol/L)
* Clinically significant (as determined by investigator) abnormalities on laboratory examination that will increase risk to the patient or interfere with data integrity
* Have any other conditions, which, in the opinion of the Investigator would make the subject unsuitable for inclusion, or could interfere with the subject participating in or completing the study
* Significant change in weight (+/- 5%) during the past month

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Change in glucose response | 2 hour
  A mixed meal tolerance test will be done to collect blood samples for glucose analysis at 0 min, 15 min, 30 min, 45 min, 60 min , 90 min and 120 min.The change in glucose response will be measured by comparing incremental area under the curve (iAUC) after ingestion of Fibre Grain meal and control Jasmine white rice meal.
Change in insulin response | 2 hour
  A mixed meal tolerance test will be done to collect blood samples for glucose analysis at 0 min, 15 min, 30 min, 45 min, 60 min , 90 min and 120 min.The change in insulin response will be measured by comparing incremental area under the curve (iAUC) after ingestion of Fibre Grain meal and control Jasmine white rice meal.

SECONDARY OUTCOMES:
Change in ghrelin level | 2 hour
  A mixed meal tolerance test will be done to collect blood samples for ghrelin analysis at 0 min, 30 min, 60 min , 90 min and 120 min.The change in ghrelin level will be measured by comparing AUC after ingestion of Fibre Grain meal and control Jasmine white rice meal.
Change in glucagon-like peptide 1 (GLP-1) level | 2 hour
  A mixed meal tolerance test will be done to collect blood samples for GLP-1 analysis at 0 min, 30 min, 60 min , 90 min and 120 min.The change in GLP-1 level will be measured by comparing AUC after ingestion of Fibre Grain meal and control Jasmine white rice meal.
Change in satiety rating | 2 hour
  A visual analogue scale (VAS) will be presented to the participants at 0, min, 30 min, 60 min , 90 min and 120 min, to indicate how they feel in response to 4 given statements by marking an "X" on a 100-mm line.
  At time T=15 min, palatability of the treatment was assessed by five characteristics, from bad (0 mm) to good (100 mm). These characteristics were visual appeal, smell, taste, texture, and overall pleasantness of the meal given. Scores were determined by measuring the distance (in mm) from the let starting point of the line to the intersection of the "X". Subjects did not discuss their ratings.The primary outcome was area under the curve (AUC) for responses on the VAS calculated using the trapezoidal rule.
Change in glucose trajectories over 14 days of continous glucose monitoring | 14 days
  FreeStyle ® Libre™ Flash glucose monitoring system (Abbott Diabetes Care, Singapore) was used for continuous glucose monitoring. During the study time frame, subjects were supplied with frozen meals for lunch and dinner to bring home. They were randomized to consumed 6 different combinations of food at 3 replacement levels for the rice: control (0%), 15% or 30% Fibre Grains. On day 14, subjects returned to the study facility to remove the flash glucose monitoring sensor and return the flash glucose monitoring reader. Subsequently, data was extracted from the reader by the study personnel. Glucose values were exported into Microsoft excel for visualization of the glucose trend over 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Mei Hui Liu, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
The plan for individual participant data will be discussed with collaborator to decide whether to be shared.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT03985566/Prot_SAP_ICF_000.pdf